CLINICAL TRIAL: NCT00005232
Title: Gubbio Study Five-year Follow-up: Lithium Countertransport, Blood Pressure, and Other Variables
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Other Study IDs: 1112; R01HL040397 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Disease

SUMMARY:
To conduct a five-year follow-up of the population of Gubbio, a town in north central Italy, in order to determine the relationship of baseline sodium-stimulated lithium countertransport to subsequent change in blood pressure and incidence of hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

The field work of the baseline or prevalence phase of the Gubbio Study on the Epidemiology of Hypertension was conducted between March 1983 and December 1985. The population sample included all individuals age 5 and over residing in the town of Gubbio. The survey involved a standardized comprehensive examination focussed on traits previously shown to be related to hypertensive and/or other adult cardiovascular diseases, and on other traits of current concern as possible risk factors. This latter category included measurement of red blood cell electrolyte concentrations and fluxes, particularly sodium-stimulated lithium countertransport. The study was planned, organized, and conducted by the Merck, Sharp and Dohme Center for Epidemiologic Research in cooperation with Gubbio civic and medical leaders, and with laboratory facilities in Gubbio, Naples, and Rome.

Follow-up examinations were conducted in the Centro di Medicina Preventiva in Gubbio which was furnished and equipped by Merck, Sharp and Dohme of Rome, Italy. Additional work was conducted at the Center for Epidemiologic Research of Merck, Sharp and Dohme in Rome, at the University of Naples, and at Northwestern University in Chicago.

DESIGN NARRATIVE:

This prospective study re-examined the 5,500 residents of Gubbio who took part in the Gubbio Population Study in 1983-1985. The data collected on follow-up focused mainly on factors related to change in blood pressure and development of hypertension and included standard physical examination, height, weight, girth, blood pressure, medical history and family medical history, urine collection for study of electrolyte excretion, venipuncture, 12-lead electrocardiogram, m-mode echocardiogram, pulse, skinfold measurement, carbon monoxide content of exhaled breath, sociodemographic data on age, marital status, education, and employment, and life style data on diet, alcohol intake, smoking, and physical activity.

Measurements made at baseline permitted assessment of whether the hypothesized positive relation of lithium countertransport to blood pressure was independent of such factors as age, sex, body mass index, alcohol intake, plasma uric acid, glucose, family history, and other variables generally associated with blood pressure. The relationship between 5-year changes in these factors, change in lithium countertransport, and in blood pressure were also examined. Several additional important unresolved questions on the epidemiology of blood pressure and hypertension were explored: the role of macronutrients and micronutrients in lithium countertransport and its change; red blood cell sodium and potassium concentrations and their relation to blood pressure; possible differences in calcium metabolism between hypertensives and normotensives; genetic polymorphisms related to lipid-lipoprotein metabolism and possible influence on blood pressure; patterns of blood pressure change in the elderly, the 639 and 341 persons age 65-74 and over 75, respectively, at baseline. Coronary heart disease incidence was also studied.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-08; Study Completion 1993-07 (Actual)

REFERENCES:
- [Background] Cirillo M, Laurenzi M. Erythrocyte and platelet volume in human hypertension. The Gubbio Study Collaborative Group. J Hypertens Suppl. 1989 Dec;7(6):S168-9. doi: 10.1097/00004872-198900076-00080. PMID 2632707
- [Background] Laurenzi M, Trevisan M. Sodium-lithium countertransport and blood pressure: the Gubbio Population Study. Hypertension. 1989 May;13(5):408-15. doi: 10.1161/01.hyp.13.5.408. PMID 2722223
- [Background] Cirillo M, Laurenzi M, Stamler J. Factors related to blood pressure in a sample of Italian children age 5 to 14: the Gubbio Population Study. Semin Nephrol. 1989 Sep;9(3):267-71. No abstract available. PMID 2781198
- [Background] Laurenzi M, Stamler R, Trevisan M, Dyer A, Stamler J. Is Italy losing the "Mediterranean advantage?" Report on the Gubbio population study: cardiovascular risk factors at baseline. Gubbio Collaborative Study Group. Prev Med. 1989 Jan;18(1):35-44. doi: 10.1016/0091-7435(89)90052-2. PMID 2710761
- [Background] Laurenzi M, Mancini M, Menotti A, Stamler J, Stamler R, Trevisan M, Zanchetti A. Multiple risk factors in hypertension: results from the Gubbio study. J Hypertens Suppl. 1990 Mar;8(1):S7-12. doi: 10.1097/00004872-199003001-00003. PMID 2332817
- [Background] Cirillo M, Laurenzi M, Trevisan M, Stamler J. Hematocrit, blood pressure, and hypertension. The Gubbio Population Study. Hypertension. 1992 Sep;20(3):319-26. doi: 10.1161/01.hyp.20.3.319. PMID 1516951
- [Background] Laurenzi M, Cirillo M, Trevisan M. The Gubbio data. Epidemiology and pathophysiology. Gubbio Study Research Group. Clin Exp Hypertens A. 1992;14(1-2):261-9. doi: 10.3109/10641969209036187. PMID 1541040
- [Background] Trevisan M, Laurenzi M. Correlates of sodium-lithium countertransport. Findings from the Gubbio Epidemiological Study. The Gubbio Collaborative Study Group. Circulation. 1991 Nov;84(5):2011-9. doi: 10.1161/01.cir.84.5.2011. PMID 1934375
- [Background] Trevisan M, Krogh V, Cirillo M, Laurenzi M, Dyer A, Stamler J. Red blood cell sodium and potassium concentration and blood pressure. The Gubbio Population Study. Ann Epidemiol. 1995 Jan;5(1):44-51. doi: 10.1016/1047-2797(94)00040-z. PMID 7728284
- [Background] Strazzullo P, Cappuccio FP. Hypertension and kidney stones: hypotheses and implications. Semin Nephrol. 1995 Nov;15(6):519-25. PMID 8588112
- [Background] Cirillo M, Laurenzi M, Panarelli W, Stamler J. Urinary sodium to potassium ratio and urinary stone disease. The Gubbio Population Study Research Group. Kidney Int. 1994 Oct;46(4):1133-9. doi: 10.1038/ki.1994.376. PMID 7861708
- [Background] Schork NJ, Weder AB, Trevisan M, Laurenzi M. The contribution of pleiotropy to blood pressure and body-mass index variation: the Gubbio Study. Am J Hum Genet. 1994 Feb;54(2):361-73. PMID 8304351
- [Background] Zanchetti A. Concepts of multiple risk factors management: the Gubbio study. J Hypertens Suppl. 1990 Mar;8(1):S3-5. doi: 10.1097/00004872-199003001-00002. PMID 2332815
- [Background] Cirillo M, Laurenzi M, Panarelli W, Trevisan M, Stamler J. Prospective analysis of traits related to 6-year change in sodium-lithium countertransport. Gubbio Population Study Research Group. Hypertension. 1999 Mar;33(3):887-93. doi: 10.1161/01.hyp.33.3.887. PMID 10082504
- [Background] Cirillo M, Senigalliesi L, Laurenzi M, Alfieri R, Stamler J, Stamler R, Panarelli W, De Santo NG. Microalbuminuria in nondiabetic adults: relation of blood pressure, body mass index, plasma cholesterol levels, and smoking: The Gubbio Population Study. Arch Intern Med. 1998 Sep 28;158(17):1933-9. doi: 10.1001/archinte.158.17.1933. PMID 9759691
- [Background] Laurenzi M, Cirillo M, Panarelli W, Trevisan M, Stamler R, Dyer AR, Stamler J. Baseline sodium-lithium countertransport and 6-year incidence of hypertension. The Gubbio Population Study. Circulation. 1997 Feb 4;95(3):581-7. doi: 10.1161/01.cir.95.3.581. PMID 9024143
- [Background] Cirillo M, Laurenzi M, Panarelli W, Trevisan M, Dyer AR, Stamler R, Stamler J. Sodium-lithium countertransport and blood pressure change over time: the Gubbio study. Hypertension. 1996 Jun;27(6):1305-11. doi: 10.1161/01.hyp.27.6.1305. PMID 8641740